CLINICAL TRIAL: NCT02649049
Title: Assessment of Dietary Intakes of Patients With Nonalcoholic Fatty Liver Disease (NAFLD)
Brief Title: Dietary Determinants in Patients With Nonalcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Type: Observational
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Associate Prof, National Nutrition and Food Technology Institute
Other Study IDs: 565
Record Dates: First submitted 2016-01-03; First posted 2016-01-07 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Dietary Intake; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Patients with NAFLD: Patients with NAFLD are the cases.
  Interventions: Other: there is no intervention
- control group: Healthy people without NAFLD are controls.
  Interventions: Other: there is no intervention

INTERVENTIONS:
Other: there is no intervention

SUMMARY:
Patients with NAFLD and matched controls will be asked about their demographic status, and their previous year dietary intakes using a validated FFQ.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18
* NAFLD was diagnosed by Fibroscan and other hepatic disorders ruled out

Exclusion Criteria:

* not completing more than 10% of the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with NAFLD diagnosed using Fibroscan without any other chronic disorders.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
nonalcoholic fatty liver disease diagnosed by Fibroscan | 6 months
  patients with confirmed diagnosis will be asked about their dietary intakes

CONTACTS AND LOCATIONS:
Locations (1):
- NNFTRI clinic, Tehran, Tehran Province, Iran